CLINICAL TRIAL: NCT02607644
Title: Clinical Evaluation of Laryngeal Tube and Laryngeal Mask Airway for Cardiac Arrest Treatment in Emergency Ambulances in Singapore
Brief Title: Laryngeal Tube vs Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Changi General Hospital (Other); KK Women's and Children's Hospital (Other Government); Ng Teng Fong General Hospital (Other); Tan Tock Seng Hospital (Other); National University Hospital, Singapore (Other); Khoo Teck Puat Hospital (Other); Singapore Civil Defence Force (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/2181
Record Dates: First submitted 2015-11-04; First posted 2015-11-18 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Cardiac Arrest
Keywords: Intubation; Ventilation; Cardiac arrest; prehospital; Laryngeal Masks; Laryngeal Tube; airway management
MeSH Terms: conditions — Heart Arrest; Respiratory Aspiration | interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laryngeal Tube (LT) (Experimental): VBM Laryngeal Tube (Intervention)
  Interventions: Device: Laryngeal Tube (LT)
- Laryngeal Mask Airway (LMA) (Active Comparator): Laryngeal Mask Airway (LMA)
  Interventions: Device: Laryngeal Mask Airway (LMA)

INTERVENTIONS:
Device: Laryngeal Mask Airway (LMA) — Laryngeal Mask Airway (LMA) for Control group
  Arms: Laryngeal Mask Airway (LMA)
Device: Laryngeal Tube (LT) — Laryngeal Tube (LT) for Intervention group
  Arms: Laryngeal Tube (LT)

SUMMARY:
Introduction: The laryngeal mask airway (LMA) is used as the primary airway by paramedics in Singapore Civil Defense Force's Emergency Ambulance Service (SCDF's EAS) in the management of out-of-hospital cardiac arrest, because endotracheal intubation requires skilled and experienced personnel, and local paramedics are not trained to this level of skill and competency. However, self-reported insertion success rates by paramedics in the field are currently only about 50-87%. Devices like the laryngeal tube have been shown to have higher placement success rates and fewer complications.

Aim: Investigators aim to evaluate the efficacy and safety of a new device, the Laryngeal Tube (LT), compared to the LMA. They hypothesize that the LT is superior to the LMA in terms of placement success rates by paramedics in SCDF's EAS, and is associated with fewer adverse events.

Methodology: Investigators propose to conduct a prospective, longitudinal multi-centre randomized trial comparing LMA and LT in patients with cardiac arrest (medical or traumatic) managed by SCDF EAS. The trial will recruit 1,015 eligible patients presenting to SCDF irrespective of destination hospital over a period of 1 year to detect an expected 15% difference in placement success rate. Currently the LMA is used as standard of care by SCDF's EAS in patients with cardiac arrest.

Results: Besides the primary outcome, the secondary outcomes of dislodgment rates, time to placement, number of attempts and adverse events will be analyzed and will be useful in guiding future SCDF cardiac arrest protocols.

DETAILED DESCRIPTION:
Endotracheal intubation (ETI) is considered the gold standard of airway management as it a definitive airway providing ventilation and prevention of aspiration in a patient unable to protect his airway. However, it can only be used by skilled, experienced personnel and can be difficult in the pre-hospital setting. It may also result in unrecognized oesophageal intubation. Currently ETI is not recommended for Singapore Civil Defence Force (SCDF) ambulances by MHA (Medical Advisory Committee) and local paramedics were not trained to this level of skill and competency. Furthermore, there has been reduced emphasis on early tracheal intubation unless achieved by highly skilled individuals to minimise interruption to chest compressions according to the 2010 resuscitation guidelines.

In view of the above reasons, ETI is not recommended by the Ministry of Home Affair's Medical Advisory Committee (MAC). Instead, the disposable laryngeal mask airway (LMA) has been used as the primary airway by paramedics in SCDF's Emergency Ambulance Service (EAS) in the management of both medical and traumatic cardiac arrest patients and is approved by the MAC for use in both adults and children.

However there can still be complications with the LMA such as incomplete seal and partial airway obstruction from mask misplacement or kinking. In addition, SCDF's self-reported success rate of LMA is only 50-87% .Hence there was a need to explore other alternatives to the LMA. The American Heart Association (AHA) recommends advanced airway adjuncts such as the Laryngeal Tube (LT) and Oesophageal-tracheal tube (Combitube) for alternative airway strategies. Other devices include the pharyngeaotracheal lumen airway and the oesophageal obdurator airway - oesophageal gastric tube airway (EOA-EGTA).

Investigators have chosen the LT as an alternative adjunct because it has a higher insertion success rate than LMA. It also has low complication such as regurgitation, vomiting and dislodgement and comes in sizes to accommodate both paediatric and adult. Method of use is quite simple as it can be inserted blindly into the oropharynx and pushed in until resistance is felt or device is fully inserted as denoted by the markings on the device.

Our long term objective is to improve existing EAS's cardiac arrest protocol and placement success rate and to lower complications and adverse events rates in out of hospital cardiac arrest. The result of the study will be reviewed by SCDF's Medical Advisory Committee (MAC). The results can also determine the choice of rescue airways used in the hospitals eg operating theatres, emergency departments, endoscopy rooms.

Primary objectives:

Investigators aim to evaluate the efficacy of the Laryngeal Tube (LT) as a primary airway in the management of cardiac arrest patients by comparing placement success rates of LT to that of LMA (Laryngeal Mask Airway) in Out-of-Hospital Cardiac Arrest managed by Singapore Civil Defence Force ambulances

Secondary Objective:

To compare the safety of the two airway devices by comparing the following outcomes:

1. Number of placement attempts required,
2. Dislodgement rates and
3. Time to successful placement of airway device.

Hypothesis:

The LT is more efficacious than the LMA as a primary airway device in the prehospital management of cardiac arrest by SCDF's EAS done by paramedics in Singapore Civil Defence Force's Emergency Ambulance Service (SCDF's EAS).

Investigators propose to conduct a prospective longitudinal multi-centre (fire stations) randomised study comparing the laryngeal mask airway (LMA) and laryngeal tube (LT ).The trial will recruit 1,015 eligible patients over 1 year. They will randomise all Emergency Ambulance Service (EAS) ambulance stations managed by SCDF into two trial groups using a longitudinal multi-centre randomised trial design. Group 1 will use new laryngeal tube (LT) protocol for 12 months and group 2 will continue laryngeal mask airway (LMA) protocol for 12 months. Investigators will record expertise/experience/training variables for each paramedic, so adjustment can be made in analysis.

Singapore General Hospital (SGH) will be submitting an ethics application to Centralised Institutional Review Board (CIRB) on behalf of SCDF to recruit all cases presenting to SCDF, irrespective of destination hospital. This is because SCDF does not have its own IRB. All the enrolled patients will be followed up by a review of their Emergency Department and hospital records for any medical related adverse effects.

The local self-reported LMA insertion success rate is 50-87%, based on a survey done as part of a larger analysis of cardiac arrest figures during the period of July 2012 to June 2013. Results from European and American airway trials involving paramedics report varying LT insertion success rates of up to 100%.

Most cardiac arrest cases occurs out-of-hospital, and most of them are conveyed by SCDF EAS. Patients will be given the treatment if all eligibility criteria are met and treatment is indicated by protocol. No written consent will be sought as this will be part of routine clinical care.

Half of the 30 SCDF ambulances will use the LT (after half day training on usage) and another half will continue with the LMA for 12 months. The treatment that each ambulance station will be providing will be randomised. Stratified randomisation with 3 strata will be carried out. The 1st strata, 2nd and 3rd stratum consist of ambulances coming from fire posts equipped with 1 ambulance, 2 ambulances and 3 ambulances respectively. Block randomisation within each stratum will be carried out to randomise the ambulances to administer LMA or LT.

Sample size calculation is based on a test for 2 proportions in a repeated measurements design. Assuming a sample size of 35 paramedics in each arm to achieve 80% power to detect an increase in successful insertion rate to 0.95 in the LT arm with 10 patient measurements per paramedic, having a Compound Symmetry covariance structure when the successful insertion proportion from the LMA arm is 0.800, the correlation between observations on the same subject is 0.5, and the alpha level is 0.05. The number of SCDF paramedics is estimated at 70, thus expect a total sample of 700 patients. Assuming a dropout rate of 45%, the investigators would need to enrol a total of 1,015 patients. This number of patients corresponds to the number of patients with out of hospital cardiac arrest (OHCA) needing intubation expected during the study period.

Frequency tables and descriptive statistics with 95% confidence intervals for all outcome variables listed above will be calculated. Associations between treatment groups and all endpoints will be analysed using the t-test/ Mann-Whitney and chi-square tests with odds ratios presented where applicable. Multivariate logistic regression will be used to adjust for relevant covariates in the analysis of primary end point of success (Y/N) of insertion.

In the control arm, the LMA will be inserted as per current SCDF protocols. The LMA can be inserted with the curved portion of the tube and the flat side of the cuff facing the patient. The patient's mouth needs to be opened and head tilted backward (except in suspected neck injury). By keeping the leading edge flat at the time of insertion, direct the cuff against the hard palate and maintain constant pressure down through the oropharynx in a smooth, continuous motion until resistance is encountered. For the intervention arm, the LT is inserted blindly into the oropharynx and pushed in until resistance is felt or device is fully inserted as denoted by the second black line. The LT has two cuffs, one at the distal and the other in the middle part of tube. The cuffs are simultaneously inflated with one syringe. The distal cuff obstructs the oesophagus and the proximal cuff occludes the pharynx. In the right position, the distal aperture should face the glottis aperture.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13-100 years old
* Cardiac arrest (medical or traumatic)
* Adjunct airway device is needed

Exclusion Criteria:

* Resuscitation is not indicated (e.g. decapitation, rigor mortis, dependant lividity)
* Pregnant women
* Conscious, intact gag reflex
* Known ingestion of caustic substances

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 965 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
successful intubation (number | 1 year
  Confirm clinically by auscultation and equal chest rise on bagging

SECONDARY OUTCOMES:
number of placement attempts required | 10 minutes
Dislodgement rates | 1 hour
Time to successful placement of airway device | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jing Chan, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore Civil Defence Force, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided